CLINICAL TRIAL: NCT05582434
Title: Factors Affecting Medication Adherence to Topical Acne Medications: a Single-center, Prospective Study Evaluating the Adherence and Patient Satisfaction to Single and Multiple Topical Acne Medications
Brief Title: Experience With Topical Acne Treatment
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00089304
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Adapalene; Gels; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- One single fixed-combination product (Experimental): Participants instructed to apply clindamycin phosphate 1.2%/adapalene 0.15%/BPO 3.1% gel once daily
  Interventions: Drug: clindamycin phosphate 1.2%/adapalene 0.15%/BPO 3.1% gel
- Two products (Experimental): Participants instructed to apply 0.3%/BPO 2.5% gel and compounded clindamycin phosphate 1.2% gel once daily
  Interventions: Drug: adapalene 0.3%/BPO 2.5% gel and compounded clindamycin phosphate 1.2% gel
- Three products (Experimental): Participants instructed to apply BPO 2.5% gel, adapalene 0.1% gel, and compounded clindamycin phosphate 1.2% gel once daily
  Interventions: Drug: Compounded BPO 2.5% gel, adapalene 0.1% gel, and compounded clindamycin phosphate 1.2% gel

INTERVENTIONS:
Drug: clindamycin phosphate 1.2%/adapalene 0.15%/BPO 3.1% gel — Single topical treatment to be applied daily to area affected once daily.
  Other Names: Cabtreo®
  Arms: One single fixed-combination product
Drug: adapalene 0.3%/BPO 2.5% gel and compounded clindamycin phosphate 1.2% gel — Two topical treatments to be applied to area affected once daily.
  Other Names: Epiduo® Forte and Clindamycin
  Arms: Two products
Drug: Compounded BPO 2.5% gel, adapalene 0.1% gel, and compounded clindamycin phosphate 1.2% gel — Three topical treatments to be applied to area affected once daily.
  Other Names: Differin®, Epsolay, Clindamycin
  Arms: Three products

SUMMARY:
Acne is a chronic condition that typically requires the use of multiple medications.1 Medication adherence is especially challenging for patients with chronic diseases and often decreases over time, especially for those using topical medications.1 Nonadherence can result in multiple negative effects including treatment failure, increased healthcare costs, and decreased quality of life. Primary nonadherence refers to problems acquiring and starting treatment. Challenges to this form of nonadherence include a lack of knowledge, misunderstanding of usage, poor communication with provider, increased cost, and fear of side effects.2 Secondary nonadherence refers to when the patient does not use the medication as prescribed. Hurdles to secondary nonadherence include delayed results, increased complexity of treatment plan, adverse effects, busy lifestyle, and inconvenience.2

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 years of age
2. Patients with a current diagnosis of acne
3. Patients who live in the US,
4. Patients have sufficient command of the English language

Exclusion Criteria:

1. Patients less than the age of 18
2. Patients without a current diagnosis of acne
3. Patients who do not live in the US
4. Patients without a sufficient command of the English language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | End of study visit - day 56
  Medication adherence measured by recording the weight of medication (in milligrams) in the bottle with electronic monitor attached
Medication Adherence | End of study visit - day 56
  Medication adherence measured by the data from the electronic monitors by frequency of use recorded by number of times opened

SECONDARY OUTCOMES:
Gender specific adherence (female subjects) | End of study visit - day 56
  Difference in medication adherence between the male and female subjects. The outcome will compare the two categories in the primary outcome
Gender specific adherence (male subjects) | End of study visit - day 56
  Difference in medication adherence between the male and female subjects. The outcome will compare the two categories in the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lott R, Taylor SL, O'Neill JL, Krowchuk DP, Feldman SR. Medication adherence among acne patients: a review. J Cosmet Dermatol. 2010 Jun;9(2):160-6. doi: 10.1111/j.1473-2165.2010.00490.x. PMID 20618564
- [Background] Moradi Tuchayi S, Alexander TM, Nadkarni A, Feldman SR. Interventions to increase adherence to acne treatment. Patient Prefer Adherence. 2016 Oct 11;10:2091-2096. doi: 10.2147/PPA.S117437. eCollection 2016. PMID 27784999
- [Background] Tan X, Al-Dabagh A, Davis SA, Lin HC, Balkrishnan R, Chang J, Feldman SR. Medication adherence, healthcare costs and utilization associated with acne drugs in Medicaid enrollees with acne vulgaris. Am J Clin Dermatol. 2013 Jun;14(3):243-51. doi: 10.1007/s40257-013-0016-x. PMID 23572294